CLINICAL TRIAL: NCT05743049
Title: Protocol to Permit Collection of Circulating Biomarkers in Pancreatic Cancer
Brief Title: Collection of Circulating Biomarkers in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 20222; 852628 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2023-02-10; First posted 2023-02-24 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood specimens: Collection of blood for analysis of various circulating biomarkers in patients with pancreatic adenocarcinoma.
  Interventions: Other: Obtaining blood for analysis of various circulating biomarkers

INTERVENTIONS:
Other: Obtaining blood for analysis of various circulating biomarkers — 4 tbsp of blood in a 1-week period, occurring no more frequently than 4 times in an 8-week period

SUMMARY:
This protocol will involve collection of blood samples from patients with a diagnosis of pancreatic adenocarcinoma for evaluation of circulating biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have a known or presumed diagnosis of pancreatic adenocarcinoma
* The subject must be a patient of the University of Pennsylvania
* The subject must be able to provide informed consent
* The subject must be 18 years of age or older

Exclusion Criteria:

. Subjects who have any clinically significant psychiatric, social, or medical condition that, in the opinion of the investigator, could increase the patient's risk, interfere with protocol adherence, or affect the patient's ability to give informed consent are ineligible to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: known or suspected diagnosis of pancreatic adenocarcinoma
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
To create a comprehensive system to collect, catalogue and store blood specimens from subjects with pancreatic cancer for future research use. | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
To create a computerized clinical data set from subjects with pancreatic cancer that contains information related to the subject's general health, disease status, treatments, and response. | Through study completion, an average of 1 year
To integrate the data and specimens to permit the most informative clinical-biologic research platform. | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark O'Hara, MD, Principal Investigator — Abramson Cancer Center, University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No